CLINICAL TRIAL: NCT02511184
Title: A PHASE 1B STUDY OF CRIZOTINIB IN COMBINATION WITH PEMBROLIZUMAB (MK-3475) IN PATIENTS WITH UNTREATED ADVANCED ALK-TRANSLOCATED NON SMALL CELL LUNG CANCER
Brief Title: Crizotinib Plus Pembrolizumab In Alk-Positive Advanced Non Small Cell Lung Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision based on the low enrollment mainly due to high efficacy drugs available in 1st line ALK-positive NSCLC (eg alectinib), not due to any safety concerns
Sponsor: Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A8081054; KEYNOTE 050 (Other: Merck Sharp & Dohme Corp); CRIZOTINIB (Other: Alias Study Number)
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-04

CONDITIONS: ALK-positive Advanced NSCLC
Keywords: crizotinib; pembrolizumab; ALK-positive NSCLC; Lung Cancer; ALK-translocated NSCLC; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Crizotinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose finding and dose expansion phases (Experimental): Find and expand the maximum tolerated dose of crizotinib in combination with pembrolizumab 200 mg iv infusion every 3 weeks.
  Interventions: Drug: Crizotinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Crizotinib — To test 3 dose levels of crizotinib in combination with pembrolizumab 200 mg iv infusion every 3 weeks
Drug: Pembrolizumab — To test pembrolizumab at 200 mg every 3 weeks in combination with crizotinib at 3 dose levels.

SUMMARY:
The purpose of this study has 2 phases, a Dose Finding Phase will determine the maximum tolerated dose . The Dose Expansion Phase will explore the safety, tolerability, and anti-tumor activity of the combination.

DETAILED DESCRIPTION:
The patients will be screened for up to 28 days before they start treatment to determine if they meet eligibility criteria. The screening procedures will include physical examination, blood work and radiological scans.

In the dose finding phase, patients who meet eligibility criteria will receive crizotinib at the dose level assigned that will be taken on daily basis and pembrolizumab 200 mg intravenous infusion every 3 weeks.

Once a Crizotinib dose level is decided, the dose expansion cohort will start enrolling patients who meet eligibility criteria.

All patients will be followed up every three weeks. Blood samples will be drawn to test for safety and tumor activities and radiological scans will be performed on certain timepoints to determine the antitumor activities.

There will be a quality of life questionnaire administered at certain time points during the study.

The study will have a quality assurance plan that addresses data validation and registry procedures. There is a plan to visit the investigator site for routine monitoring and auditing.

The team will conduct source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (e.g., medical records, paper or electronic case report forms, or interactive voice response systems).

The study will also include a statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives of this study, as specified in the study protocol or statistical plan.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proved diagnosis of locally advanced recurrent or metastatic non-squamous NSCLC that is not suitable for local curative treatment.
* Alk-positive NSCLC as determined by a test that is approved or validated for use as a companion diagnostic test.
* No prior systemic therapy for metastatic disease.
* Adjuvant chemotherapy more than 12 months prior to study enrollment.
* Measurable disease as per RECIST 1.1
* ECOG PS 0 or 1.

Exclusion Criteria:

* Prior exposure to ALK receptor tyrosine kinase inhibitor, anti-PD1, anti-PDL1 or any drug targeting T-cell checkpoint pathways.
* known diagnosis of immunodeficiency or is receiving systemic steroid therapy or other form of immunosuppressive therapy within 7 days of clinical trial treatment.
* Active autoimmune disease that has required systemic treatment in the past 3 months.
* History of extensive disseminated interstitial fibrosis or any grade of interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, IDS Pharmacy, Birmingham, Alabama
  - City of Hope National Medical Center, Duarte, California
  - UC San Diego Moores Cancer Center - Investigational Drug Services, La Jolla, California
  - UC San Diego Medical Center - La Jolla(Thornton Hospital), La Jolla, California
  - University Of California / San Diego Moores Cancer Center, La Jolla, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Investigational Drug Services Pharmacy, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8081054&StudyName=A%20Phase%201b%20Study%20Of%20Crizotinib%20In%20Combination%20With%20Pembrolizumab%20%28mk-3475%29%20In%20Patients%20With%20Untreated%20Advanced%20Alk-translocated%20Non%20Small%20Cell%20Lung%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib + Pembrolizumab: Participants were administered combination therapy of crizotinib (250 mg capsule orally, twice daily) and pembrolizumab (200 mg via 30-minute intravenous infusion, every 3 weeks) until disease progression and no clinical benefit, or unacceptable toxicity, death, or consent withdrawal, whichever occurred first.
- Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab: Participants were administered monotherapy of crizotinib (250 mg capsule orally, twice daily) for 3 weeks, and if tolerated, followed by combination therapy of crizotinib (250 mg capsule orally, twice daily) and pembrolizumab (200 mg via 30-minute intravenous infusion, every 3 weeks) until disease progression and no clinical benefit, or unacceptable toxicity, death, or consent withdrawal, whichever occurred first.
Period: Overall Study
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Started | 2 | 7
Completed | 0 | 0
Not Completed | 2 | 7
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study terminated by sponsor | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants enrolled in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab | Total
Number analyzed (Participants) | 2 | 7 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (12) | 56.4 (13) | 58.2 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 5 | 7
  Asian | 0 | 1 | 1
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT)
Description: Dose-limiting toxicity (DLT) was defined as any of the following adverse events (AEs) occurring in the first 2 cycles of treatment (6 weeks) which were attributable to crizotinib, pembrolizumab or both: hematologic toxicities including Grade 4 neutropenia, febrile neutropenia, Grade greater than or equal to (>=) 3 neutropenic infection, Grade >=3 thrombocytopenia with bleeding; Grade 4 thrombocytopenia; non-hematologic toxicities including Grade >=3 toxicities (non-laboratory), Grade >=3 nausea, vomiting, or diarrhea despite maximal therapy, non-hematologic Grade >=3 laboratory value if medical intervention was required to treat the participant or the abnormality led to hospitalization; inability to complete at least 80 percent of the first 2-cycle doses of crizotinib or both infusions of pembrolizumab within the DLT observation period due to treatment-related toxicity. Grade was based on National Cancer Institute Common Terminology Criteria for AEs (NCI CTCAE) version 4.03.
Time Frame: 6 weeks
Population: DLT evaluable population included all participants enrolled in the Dose Finding Phase who received at least 1 dose of crizotinib or pembrolizumab, and either experienced DLT during the first 2 cycles, or completed the observation period for the first 2 cycles of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
Participants | 2 | 2

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events
Description: AE was defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of the causal relationship to study treatment. Treatment-emergent AEs (TEAEs) were defined as AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Causality to study treatment was determined by the investigator. Severity was graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 2 years
Population: The safety analysis set included all enrolled participants who received at least 1 dose of crizotinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
Participants
  All-causality AE | 2 | 7
  All-causality SAE | 2 | 1
  Crizotinib-related AE | 2 | 7
  Crizotinib-related SAE | 0 | 0
  Pembrolizumab-related AE | 2 | 6
  Pembrolizumab-related SAE | 2 | 1
  Grade 1 all-causality AE | 0 | 1
  Grade 2 all-causality AE | 0 | 2
  Grade 3 all-causality AE | 0 | 4
  Grade 4 all-causality AE | 1 | 0
  Grade 5 all-causality AE | 1 | 0

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR refers to percentage of participants who achieved complete response (CR) or partial response (PR) in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1. A participant achieved CR if both target and non-target lesions achieved CR, no new lesions; achieved PR if target lesions achieved CR or PR, non-target lesions were assessed as non-CR/non-progressive disease (PD) or not evaluated, and no new lesions. For target lesions, CR: complete disappearance of all target lesions; PR: >= 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. For non-target lesions, CR: disappearance of all non-target lesions and normalization of tumor marker levels and all lymph nodes must be non-pathological in size; non-CR/non-PD: persistence of any non-target lesions and/or tumor marker level above the normal limits.
Time Frame: Baseline, Week 9 and every 6 weeks thereafter, for about 2 years
Population: The analysis population included all treated participants who had an adequate baseline tumor assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
percentage of participants | 50 | 57.1

4. Secondary Outcome: Duration of Response
Description: Duration of Response (DR) was defined as the time from first documentation of objective tumor response (CR or PR) that was subsequently confirmed, to the first documentation of objective tumor progression or to death on study due to any cause, whichever occurred first.
Time Frame: Baseline, Week 9 and every 6 weeks thereafter, for about 2 years
Population: The analysis population included all participants who achieved complete response or partial response.
Measure: Median (Full Range); unit: days
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 1 | 4
days | 85 [85 to 85] | 242 [126 to 339]

5. Secondary Outcome: Time to Tumor Response
Description: Time to Tumor Response (TTR) was defined as the time from the first dose of crizotinib or pembrolizumab to the first documentation of objective tumor response (CR or PR) that was subsequently confirmed.
Time Frame: Baseline, Week 9 and every 6 weeks thereafter, for about 2 years
Population: The analysis population included all participants who achieved complete response or partial response.
Measure: Median (Full Range); unit: days
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 1 | 4
days | 57 [57 to 57] | 83 [77 to 87]

6. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) was defined as the time from the first dose of crizotinib or pembrolizumab to the first documentation of objective tumor progression or death on-study due to any cause, whichever occurred first. For participants who did not have documented objective progression during the study or were alive at last contact, the date of last contact was used.
Time Frame: Baseline, Week 9 and every 6 weeks thereafter, for about 2 years
Population: The analysis population included all treated participants who had an adequate baseline tumor assessment.
Measure: Median (Full Range); unit: days
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
days | 131.5 [122 to 141] | 211 [1 to 418]

7. Secondary Outcome: 6-Month, 12-Month and 18-Month Progression Free Survival Probabilities
Description: PFS probabilities were defined as the probability of being alive and progression free at 6, 12 and 18 months after the date of first dose based on the Kaplan Meier estimate.
Time Frame: Month 6, Month 12, and Month 18
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) was defined as the time from the first dose of crizotinib or pembrolizumab to the date of death due to any cause. For participants who were alive at last contact, the date of last contact was used.
Time Frame: Day 1 to end of study (for about 2 years)
Population: The analysis population included all treated participants who had an adequate baseline tumor assessment.
Measure: Median (Full Range); unit: days
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
days | 452.5 [122 to 783] | 428 [272 to 730]

9. Secondary Outcome: 12-Month and 18-Month Overall Survival Probabilities
Description: OS probabilities were defined as the probability of being alive at 12 and 18 months after the date of first dose based on the Kaplan Meier estimate.
Time Frame: Month 12 and Month 18
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Maximum Grade in Laboratory Hematology Test Shifting From Grade 0, 1 or 2 at Baseline to Grade 3 or 4 During Treatment
Description: Hematology evaluation included hemoglobin, platelets, white blood cell, absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils, and absolute basophils. Hematology test results were graded by NCI CTCAE version 4.03.
Time Frame: 2 years
Population: The safety analysis set included all enrolled participants who received at least 1 dose of crizotinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
Participants
  Anemia | 0 | 0
  Hemoglobin increased | 0 | 0
  Lymphocyte count increased | 0 | 0
  Lymphopenia | 0 | 2
  Absolute neutrophils | 0 | 0
  platelets | 0 | 0
  White blood cells | 0 | 0

11. Secondary Outcome: Number of Participants With Maximum Grade in Laboratory Chemistry Test Shifting From Grade 0, 1 or 2 at Baseline to Grade 3 or 4 During Treatment
Description: Chemistry evaluation included alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, sodium, potassium, magnesium, chloride, total calcium, total bilirubin, blood urea nitrogen or urea, creatinine, uric acid, glucose, albumin, phosphorous or phosphate, thyroid function tests including thyroid-stimulating hormone, T3 and free T4. Chemistry test results were graded by NCI CTCAE version 4.03.
Time Frame: 2 years
Population: The safety analysis set included all enrolled participants who received at least 1 dose of crizotinib or pembrolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
Participants
  Alanine aminotransferase | 1 | 3
  Alkaline phosphatase | 0 | 0
  Aspartate aminotransferase | 1 | 1
  Total bilirubin | 0 | 0
  Creatine kinase: number analyzed (Participants) | 1 | 0
  Creatine kinase | 0 | 0
  Creatinine | 0 | 0
  Gamma-glutamyl transferase: number analyzed (Participants) | 1 | 0
  Gamma-glutamyl transferase | 0 | 0
  Hypercalcemia | 0 | 0
  Hyperglycemia | 0 | 1
  Hyperkalemia | 0 | 0
  Hypermagnesemia | 0 | 0
  Hypernatremia | 0 | 0
  Hypoalbuminemia | 0 | 0
  Hypocalcemia | 0 | 0
  Hypoglycemia | 0 | 0
  Hypokalemia | 0 | 0
  Hypomagnesemia | 0 | 0
  Hyponatremia | 1 | 1
  Hypophosphatemia | 0 | 1

12. Secondary Outcome: Plasma Concentration Summary of Crizotinib for "Crizotinib + Pembrolizumab" Group
Time Frame: Prior to crizotinib morning dose on Day 1 of Cycles 1, 2, 4, 6, and 8, and at the End of Treatment visit (28 to 35 days after the last dose of study treatment)
Population: The analysis population included all treated participants who had at least 1 crizotinib concentration measurement.
Measure: Median (Full Range); unit: nanograms/milliliter (ng/mL)
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2
nanograms/milliliter (ng/mL)
  Day 1 of Cycle 1: pre-dose | 0 [0 to 0]
  Day 1 of Cycle 2: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 2: pre-dose | 379 [379 to 379]
  Day 1 of Cycle 4: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 4: pre-dose | 147 [147 to 147]
  Day 1 of Cycle 6: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 6: pre-dose | 235 [235 to 235]
  Day 1 of Cycle 8: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 8: pre-dose | 257 [257 to 257]
  End of treatment | 166.04 [8.08 to 324]

13. Secondary Outcome: Plasma Concentration Summary of Crizotinib for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Time Frame: Pre-dose, and 1, 2, 4, 6 and 8 hours post-dose on Day 15 of monotherapy and on Day 1 of Cycle 6; prior to crizotinib morning dose on Day 1 of Cycles 1, 2, 4, 6, and 8, and at the End of Treatment visit (28-35 days after the last dose of study treatment)
Population: The analysis population included all treated participants who had at least 1 crizotinib concentration measurement.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 7
ng/mL
  Day 15 of monotherapy: pre-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: pre-dose | 273 [79.9 to 531]
  Day 15 of monotherapy: 1 hour post-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 1 hour post-dose | 262.5 [191 to 300]
  Day 15 of monotherapy: 2 hours post-dose | 345 [159 to 455]
  Day 15 of monotherapy: 4 hours post-dose | 331 [133 to 375]
  Day 15 of monotherapy: 6 hours post-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 6 hours post-dose | 278 [115 to 373]
  Day 15 of monotherapy: 8 hours post-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 8 hours post-dose | 294.5 [129 to 382]
  Day 1 of Cycle 1: pre-dose: number analyzed (Participants) | 6
  Day 1 of Cycle 1: pre-dose | 272.5 [176 to 337]
  Day 1 of Cycle 2: pre-dose | 131 [0.842 to 249]
  Day 1 of Cycle 4: pre-dose: number analyzed (Participants) | 6
  Day 1 of Cycle 4: pre-dose | 194.5 [37.5 to 352]
  Day 1 of Cycle 6: pre-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: pre-dose | 249 [175 to 311]
  Day 1 of Cycle 6: 1 hour post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 1 hour post-dose | 272 [184 to 281]
  Day 1 of Cycle 6: 2 hours post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 2 hours post-dose | 274 [194 to 497]
  Day 1 of Cycle 6: 4 hours post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 4 hours post-dose | 317 [198 to 450]
  Day 1 of Cycle 6: 6 hours post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 6 hours post-dose | 301 [172 to 369]
  Day 1 of Cycle 6: 8 hours post-dose: number analyzed (Participants) | 4
  Day 1 of Cycle 6: 8 hours post-dose | 229.5 [173 to 367]
  Day 1 of Cycle 8: pre-dose: number analyzed (Participants) | 4
  Day 1 of Cycle 8: pre-dose | 244.5 [159 to 285]
  End of treatment: number analyzed (Participants) | 4
  End of treatment | 24.65 [0.65 to 489]

14. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Crizotinib for "Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 12
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

15. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Crizotinib for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 13
Population: Data were not collected.
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

16. Secondary Outcome: Area Under the Plasma Concentration Time Curve From 0 to 8 Hours (AUC0-8) of Crizotinib for "Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 12
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

17. Secondary Outcome: Area Under the Plasma Concentration Time Curve From 0 to 8 Hours (AUC0-8) of Crizotinib for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 13
Population: Data were not collected.
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

18. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUCtau) of Crizotinib for "Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 12
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

19. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUCtau) of Crizotinib for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 13
Population: Data were not collected.
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

20. Secondary Outcome: Apparent Plasma Clearance (CL/F) of Crizotinib for "Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 12
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

21. Secondary Outcome: Apparent Plasma Clearance (CL/F) of Crizotinib for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Time Frame: as for outcome 13
Population: Data were not collected.
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

22. Secondary Outcome: Plasma Concentration Summary of PF-06260182 for "Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 12
Population: The analysis population included all treated participants who had at least 1 PF-06260182 concentration measurement.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2
ng/mL
  Day 1 of Cycle 1: pre-dose | 0 [0 to 0]
  Day 1 of Cycle 2: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 2: pre-dose | 182 [182 to 182]
  Day 1 of Cycle 4: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 4: pre-dose | 46.4 [46.4 to 46.4]
  Day 1 of Cycle 6: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 6: pre-dose | 99.1 [99.1 to 99.1]
  Day 1 of Cycle 8: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 8: pre-dose | 67 [67 to 67]
  End of treatment | 56.58 [2.16 to 111]

23. Secondary Outcome: Plasma Concentration Summary of PF-06260182 for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 13
Population: The analysis population included all treated participants who had at least 1 PF-06260182 concentration measurement.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 7
ng/mL
  Day 15 of monotherapy: pre-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: pre-dose | 91.35 [28.4 to 148]
  Day 15 of monotherapy: 1 hour post-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 1 hour post-dose | 74.15 [46.8 to 93.9]
  Day 15 of monotherapy: 2 hours post-dose | 84.3 [52.3 to 141]
  Day 15 of monotherapy: 4 hours post-dose | 107 [53.3 to 117]
  Day 15 of monotherapy: 6 hours post-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 6 hours post-dose | 91.85 [45.8 to 105]
  Day 15 of monotherapy: 8 hours post-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 8 hours post-dose | 84.5 [42.5 to 129]
  Day 1 of Cycle 1: pre-dose: number analyzed (Participants) | 6
  Day 1 of Cycle 1: pre-dose | 83.2 [40.3 to 107]
  Day 1 of Cycle 2: pre-dose | 21.6 [0 to 65.1]
  Day 1 of Cycle 4: pre-dose: number analyzed (Participants) | 6
  Day 1 of Cycle 4: pre-dose | 61.3 [8.55 to 98.3]
  Day 1 of Cycle 6: pre-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: pre-dose | 74.5 [30.1 to 94.1]
  Day 1 of Cycle 6: 1 hour post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 1 hour post-dose | 69.8 [30.8 to 80.6]
  Day 1 of Cycle 6: 2 hours post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 2 hours post-dose | 65.8 [40.8 to 144]
  Day 1 of Cycle 6: 4 hours post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 4 hours post-dose | 73.3 [31.4 to 158]
  Day 1 of Cycle 6: 6 hours post-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 6 hours post-dose | 77.7 [38.2 to 139]
  Day 1 of Cycle 6: 8 hours post-dose: number analyzed (Participants) | 4
  Day 1 of Cycle 6: 8 hours post-dose | 60.6 [38.4 to 111]
  Day 1 of Cycle 8: pre-dose: number analyzed (Participants) | 4
  Day 1 of Cycle 8: pre-dose | 62.75 [32.1 to 83.9]
  End of treatment: number analyzed (Participants) | 4
  End of treatment | 2.75 [0 to 112]

24. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of PF-06260182 for "Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 12
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

25. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of PF-06260182 for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 13
Population: Data were not collected.
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

26. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUCtau) of PF-06260182 for "Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 12
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

27. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over the Dosing Interval (AUCtau) of PF-06260182 for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 13
Population: Data were not collected.
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

28. Secondary Outcome: Metabolite (PF-06260182) to Parent (Crizotinib) AUCtau Ratio for "Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 12
Population: Data were not collected.
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

29. Secondary Outcome: Metabolite (PF-06260182) to Parent (Crizotinib) AUCtau Ratio for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 13
Population: Data were not collected.
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 0

30. Secondary Outcome: Metabolite (PF-06260182) to Parent (Crizotinib) Concentration Ratio for "Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 12
Population: The analysis population included all treated participants who had at least 1 PF-06260182 concentration measurement and at least 1 crizotinib concentration measurement.
Measure: Median (Full Range); unit: ratio
Arm/Group | Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2
ratio
  Day 1 of Cycle 1: pre-dose: number analyzed (Participants) | 0
  Day 1 of Cycle 2: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 2: pre-dose | 0.480 [0.480 to 0.480]
  Day 1 of Cycle 4: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 4: pre-dose | 0.316 [0.316 to 0.316]
  Day 1 of Cycle 6: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 6: pre-dose | 0.422 [0.422 to 0.422]
  Day 1 of Cycle 8: pre-dose: number analyzed (Participants) | 1
  Day 1 of Cycle 8: pre-dose | 0.261 [0.261 to 0.261]
  End of treatment | 0.305 [0.267 to 0.343]

31. Secondary Outcome: Metabolite (PF-06260182) to Parent (Crizotinib) Concentration Ratio for "Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab" Group
Description: PF-06260182 is a metabolite of crizotinib.
Time Frame: as for outcome 13
Population: The analysis population included all participants who had at least 1 PF-06260182 concentration measurement and at least 1 crizotinib concentration measurement.
Measure: Median (Full Range); unit: ratio
Arm/Group | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 7
ratio
  Day 15 of monotherapy: pre-dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: pre-dose | 0.334 [0.274 to 0.401]
  Day 15 of monotherapy: 1 hour post dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 1 hour post dose | 0.275 [0.226 to 0.367]
  Day 15 of monotherapy: 2 hours post dose | 0.307 [0.185 to 0.365]
  Day 15 of monotherapy: 4 hours post dose | 0.321 [0.275 to 0.401]
  Day 15 of monotherapy: 6 hours post dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 6 hours post dose | 0.330 [0.268 to 0.398]
  Day 15 of monotherapy: 8 hours post dose: number analyzed (Participants) | 6
  Day 15 of monotherapy: 8 hours post dose | 0.311 [0.263 to 0.338]
  Day 1 of Cycle 1: pre-dose: number analyzed (Participants) | 6
  Day 1 of Cycle 1: pre-dose | 0.311 [0.229 to 0.376]
  Day 1 of Cycle 2: pre-dose | 0.217 [0 to 0.303]
  Day 1 of Cycle 4: pre-dose: number analyzed (Participants) | 6
  Day 1 of Cycle 4: pre-dose | 0.293 [0.228 to 0.355]
  Day 1 of Cycle 6: pre-dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: pre-dose | 0.258 [0.172 to 0.361]
  Day 1 of Cycle 6: 1 hour post dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 1 hour post dose | 0.249 [0.145 to 0.287]
  Day 1 of Cycle 6: 2 hours post dose | 0.239 [0.210 to 0.290]
  Day 1 of Cycle 6: 4 hours post dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 4 hours post dose | 0.231 [0.159 to 0.351]
  Day 1 of Cycle 6: 6 hours post dose: number analyzed (Participants) | 5
  Day 1 of Cycle 6: 6 hours post dose | 0.258 [0.219 to 0.406]
  Day 1 of Cycle 6: 8 hours post dose: number analyzed (Participants) | 4
  Day 1 of Cycle 6: 8 hours post dose | 0.264 [0.212 to 0.302]
  Day 1 of Cycle 8: pre-dose: number analyzed (Participants) | 4
  Day 1 of Cycle 8: pre-dose | 0.244 [0.202 to 0.323]
  End of treatment: number analyzed (Participants) | 4
  End of treatment | 0.105 [0 to 0.229]

32. Secondary Outcome: Serum Concentration of Pembrolizumab
Time Frame: Prior to and at end of pembrolizumab infusion, 120 hours and 336 hours post Day 1 dosing of Cycle 1; pre-dose on Day 1 of Cycles 2, 4,6, 8, 12 and 16; end of Day 1 dosing of Cycle 8; End of Treatment visit
Population: The analysis population included all treated participants who had at least 1 pembrolizumab concentration measurement.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 7
ng/mL
  Day 1 of Cycle 1: pre-dose | 0 [0 to 0] | 0 [0 to 0]
  Day 1 of Cycle 1: end of infusion: number analyzed (Participants) | 2 | 5
  Day 1 of Cycle 1: end of infusion | 63150 [38300 to 88000] | 61400 [34600 to 102000]
  Day 8 of Cycle 1: 120 hours post Day 1 dosing | 25550 [20600 to 30500] | 26800 [19100 to 31900]
  Day 15 of Cycle 1: 336 hours post Day 1 dosing | 19600 [14800 to 24400] | 20100 [11000 to 23700]
  Day 1 of Cycle 2: pre-dose: number analyzed (Participants) | 2 | 6
  Day 1 of Cycle 2: pre-dose | 9840 [8680 to 11000] | 15750 [8020 to 19600]
  Day 1 of Cycle 4: pre-dose: number analyzed (Participants) | 0 | 5
  Day 1 of Cycle 4: pre-dose |  | 31600 [18200 to 37300]
  Day 1 of Cycle 6: pre-dose: number analyzed (Participants) | 0 | 4
  Day 1 of Cycle 6: pre-dose |  | 37000 [28500 to 64000]
  Day 1 of Cycle 8: pre-dose: number analyzed (Participants) | 0 | 4
  Day 1 of Cycle 8: pre-dose |  | 38800 [26600 to 64500]
  Day 1 of Cycle 8: end of infusion: number analyzed (Participants) | 0 | 3
  Day 1 of Cycle 8: end of infusion |  | 14300 [11700 to 14500]
  Day 1 of Cycle 12: pre-dose: number analyzed (Participants) | 0 | 2
  Day 1 of Cycle 12: pre-dose |  | 99350 [85700 to 113000]
  Day 1 of Cycle 16: pre-dose: number analyzed (Participants) | 0 | 1
  Day 1 of Cycle 16: pre-dose |  | 29300 [29300 to 29300]
  End of treatment: number analyzed (Participants) | 1 | 5
  End of treatment | 10800 [10800 to 10800] | 27500 [3370 to 45800]

33. Secondary Outcome: Number of Participants With Programmed Death Receptor-1 Ligand-1 (PD-L1) Expression Level Meeting Pre-defined Criteria
Description: Archived formalin-fixed, paraffin-embedded tumor issue block was collected at screening. PD-L1 assessment was performed using immunohistochemistry. A sample was considered negative if tumor proportion score was less than 1%; positive if tumor proportion score was greater than or equal to 1%; strong positive if tumor proportion score was greater than or equal to 50%.
Time Frame: Screening
Population: The analysis population included all participants who had evaluable PD-L1 measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
Number analyzed (Participants) | 2 | 6
Participants
  Negative | 1 | 1
  Positive | 1 | 3
  Strong positive | 0 | 2

ADVERSE EVENTS:
Time Frame: 2 years
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and nonserious in another participant, or one participant may have experienced both serious and nonserious event during study.
Arm/Group | Crizotinib + Pembrolizumab | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/2 | 1/7
Other Adverse Events (participants affected / at risk) | 2/2 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crizotinib + Pembrolizumab (N=2) | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab (N=7)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Crizotinib + Pembrolizumab (N=2) | Crizotinib Monotherapy Followed by Crizotinib + Pembrolizumab (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (4) | 5 (8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3) | 5 (7)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (2) | 2 (2)
Fatigue (General disorders) | 1 (5) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (5) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (7) | 6 (12)
Aspartate aminotransferase increased (Investigations) | 2 (6) | 5 (8)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 3 (3)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (4)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (2) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (7)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Some of the pre-defined outcome measures could not be analyzed because of premature termination, which was based on low enrollment rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT02511184/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT02511184/SAP_001.pdf